CLINICAL TRIAL: NCT06721026
Title: Re-evaluation of the Muscle-full Effect During Continuously Elevated Amino Acid Availability in Healthy Young Males
Acronym: Muscle-full
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC24-028
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Muscle Protein Synthesis
Keywords: amino acid infusion; tracer methodology; muscle biopsy

STUDY DESIGN:
Intervention Model Description: Cross-sectional, non-therapeutic, intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous amino acid infusion (Experimental): Tracer infusions combined with infusion of a mixture of amino acids
  Interventions: Other: Continuous intravenous stable isotope amino acid tracer infusion; Other: Amino acid infusion

INTERVENTIONS:
Other: Continuous intravenous stable isotope amino acid tracer infusion — During the single 12 h trial day, a primed continuous stable isotope infusion will run in order to assess muscle protein synthesis in the basal (4 h) and post-prandial (8 h) state.
Other: Amino acid infusion — In order to assess muscle protein synthesis rates during continuous elevated plasma amino acid availability, the amino acid infusion solution Vamin®14 EF will be used. Vamin® 14EF contains 85g amino acids per liter and will be administered in the post-prandial period for 8 hours to ensure a constant rate of amino acid infusion over the full assessment period of the primary outcome measure.

SUMMARY:
Muscle tissue consists of proteins. These proteins are built up of a collection of smaller building blocks: amino acids. When protein is consumed, it gets digested and absorbed into the blood. The body can use these amino acids, by taking them up from thecirculation. By consuming sufficient protein through our diet, we ensure that the body is provided with enough amino acids to enable muscle protein building. Sufficient muscle protein synthesis is important for maintaining muscle function and strength.

Previous research has shown that when 20 to 25g of protein is eaten, muscle protein synthesis is maximized. It is therefore recommended to eat 20g of protein per meal. However, it is currently unclear what happens to muscle protein synthesis rates if multiple meals are eaten. When multiple meals are consumed, amino acids appear in the circulation for prolonged period of time.

Theoretically, when there are a high amino acid concentrations in the blood, muscle protein synthesis rates will increase. Contrary to this theory, a study more than 20 years ago showed otherwise. It was observed that muscle protein synthesis rates are only elevated for2 hours afterwhich they decrease again. This phenomenon was referred to as the "muscle-full" effect. Because this phenomenon is in contrast with more previous studies, the objective is to replicate that study. This is important so that nutritional advice for healthy, but also clinical populations in the future can be improved.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Aged between 18 - 35 years
* Healthy (assessed based on routine medical questionnaire)
* BMI between 18.5 - 30 kg/m2

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Smoking
* Involved in progressive exercise training
* A history of neuromuscular problems
* Use of anticoagulants
* Recent (<12 months) participation in amino acid tracer (L-[ring-13C6] phenylalanineand L-[3,5-2H2]-tyrosine) studies
* Use of medication known to affect (muscle) protein metabolism (e.g. corticosteroids, non-steroidal anti-inflammatory drugs, acne medication)
* Phenylketonuria
* Diagnosed with or history of liver damage
* Diagnosed with or history of severe kidney damage and/or malfunction
* Diagnosed with inability to break down amino acids

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis during continuous elevated plasma amino acid avaialbility in healthy young males | 8 hours
  The primary endpoint is muscle protein synthesis rates (in %/h) over the full assessment period (8 h) as determined with contemporary stable isotope tracer methodology combined with repeated blood and muscle sampling. Muscle protein synthesis are calculated using plasma as precursor pool and the tracer enrichment in the muscle (measured with UPLC and GC-IRMS).

SECONDARY OUTCOMES:
Basal muscle protein synthesis rates | 3 hours
  Basal muscle protein synthesis rates (in %/h) will be assessed over a 3h period as determined with contemporary stable isotope tracer methodology combined with repeated blood and muscle sampling. Muscle protein synthesis are calculated using plasma as precursor pool and the tracer enrichment in the muscle biopsy (measured with UPLC and GC-IRMS).
Whole-body protein kinetics | 8 hours
  Including total rate of appearance, exogenous rate of appearance, endogenous rate of appearance, rate of disappearance based (all expressed as μmol/kg/min) on tracer plasma amino acid concentrations over time (measured with UPLC)
Whole-body protein metabolism | 8 hours
  synthesis, breakdown, oxidation, net balance (all expressed as μmol/kg/h). Based on amino acid concentrations in plasma and breath samples (measured with UPLC and GC-IRMS).

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request